CLINICAL TRIAL: NCT04543162
Title: Usefulness of Biomarkers in the Management of Mild Traumatic Brain Injury in Adults
Brief Title: Usefulness of Biomarkers in the Management of Mild Traumatic Brain Injury in Adults (Biotraumap)
Acronym: Biotraumap
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 BOUVIER (Biotraumap); 2019-A01228-49 (Other: ANSM)
Record Dates: First submitted 2019-09-26; First posted 2020-09-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury; Intracranial Injury
Keywords: Glasgow Coma Scale (GCS) score of 15; S100B; Mild Traumatic Brain Injury; Brain biomarkers; Cerebral biomarkers; Intracranial lesions
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Collection of additional blood volume (approximately 7 mL) during blood tests provided as part of the usual medical care in emergencies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Mild Traumatic Brain Injury: patients with Mild Traumatic Brain Injury

SUMMARY:
The indication of cranial computed tomography (CCT) is difficult to define for patients with mild traumatic brain injury (mTBI). For mTBI patients with a medium risk of intracranial complications, CCT scans are indicated although 90% of them are normal.

The interest of the S100B protein has been widely demonstrated in the management of mTBI in adults. Its serum concentration (for blood sampling drawn less than 3 hours after trauma) can accurately predict a normal CCT scan for mTBI patients with a medium risk of intracranial complications. That's why, serum assay of the S100B protein is routinely used in the Emergency Department of Clermont-Ferrand University Hospital for the treatment of patients with mTBI.

The objective of the study is to optimize the management strategy for mTBI patients by blood testing of new brain biomarkers. These biomarkers are synthesized by brain cells and are released into the blood in case of intracranial lesions.

DETAILED DESCRIPTION:
Other biomarkers of brain damage, involved in the pathophysiology of head trauma, are also known. These are, for example, GFAP (Glial Fibrillary Acidic Protein), UCH-L1 (Ubiquitine Carboxy Terminal Hydrolase L1), NSE (Neurone Specific Enolase), Tau, SBDP (Spectrin Breakdown Products) or NFL (Neurofilament) protein. To date, the too limited number of studies doesn't enable the use of these biomarkers routinely. Therefore we will study the interest of these biomarkers in the management of adult patients' mTBI. We wish to set a collection of biological samples drawn from 1500 patients consulting for mTBI (with a medium risk of intracranial complications) at the Emergency Department of Clermont-Ferrand University Hospital, and requiring an assay of the S100B protein.

The study will take place over a period of 36 months at Clermont-Ferrand University Hospital. Patients cared for mTBI when they come to the Emergency Department will be recruited according to the inclusion criteria. In case of no opposition, when having their blood drawn, one more tube will be drawn per patient. Then, the obtained serum will be frozen at -80 ° C for the next assays of the cerebral biomarkers such as: GFAP, UCH-L1, NSE, Tau, SBDP, NFL, etc. A later 2-weeks' telephone call after the head trauma will be made by a member of the staff of the Department of Biochemistry and Molecular Genetics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient, major
* Patient admitted to the Emergency Department for mTBI, with a medium risk of intracranial lesions according to the SFMU (French Emergency Medicine Society) criteria, for which an S100B protein assay is indicated:
* GCS score of 15 with at least one associated risk factor: amnesia facts more than 30 minutes before the mTBI loss of consciousness, anti platelet aggregating agent
* Time between mTBI and blood draw (for the S100B protein assay) less than 3 hours.
* Patient covered by a Social Security scheme.

Exclusion Criteria:

* Patient classified in the high risk group of intracranial lesions according to SFMU criteria :
* GCS score less than 15, 2 hours after the trauma
* Focused neurological deficit
* Post-traumatic convulsion
* Suspicion of open fracture of the skull or embarrassment
* Any sign of fracture of the base of the skull (hemotympanum, bilateral periorbital bruise, otorrhea or rhinorrhea of cerebrospinal fluid)
* Treatment with anticoagulants
* More than one episode of vomiting.
* Patient classified in the group at low risk of intracranial lesions according to the SFMU criteria, presenting a GCS score of 15 without any criteria for moderate or high risk groups of intracranial lesions.
* Patient consulting for moderate or severe head trauma (GCS score less than 13).
* Refusal of the patient (signature of the opposition form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild Traumatic Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of cerebral biomarkers GFAP | Day 0
  Evaluate the diagnostic value of cerebral biomarkers GFAP (ng/L)
Diagnostic value of cerebral biomarkers UCH-L1 | Day 0
  Evaluate the diagnostic value of cerebral biomarkers UCH-L1 (ng/L)
Diagnostic value of cerebral biomarkers NSE | Day 0
  Evaluate the diagnostic value of cerebral biomarkers NSE (µg/L)
Diagnostic value of cerebral biomarkers Tau | Day 0
  Evaluate the diagnostic value of cerebral biomarkers TAU (ng/L)
Diagnostic value of cerebral biomarkers SBDP | Day 0
  Evaluate the diagnostic value of cerebral biomarkers SBDP (µg/L)
Diagnostic value of cerebral biomarkers NFL | Day 0
  Evaluate the diagnostic value of cerebral biomarkers NFL (ng/L)

SECONDARY OUTCOMES:
Utility of serum biomarker measurement with respect to reduction of the cost of management | Day 0
  Calculate this cost reduction compared to the cost of a cerebral tomodensitometry
Risk factors (antiplatelet agent) on biomarker results | Day 0
  Collect information from medical records and assess the impact on biomarker results from statistical tests
risk factors (loss of consciousness) on biomarker results | Day 0
  Collect information from medical records and assess the impact on biomarker results from statistical tests
risk factors (amnesia) on biomarker results | Day 0
  Collect information from medical records and assess the impact on biomarker results from statistical tests

CONTACTS AND LOCATIONS:
Overall Officials: Damien Bouvier, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Allouchery G, Moustafa F, Roubin J, Pereira B, Schmidt J, Raconnat J, Pic D, Sapin V, Bouvier D. Clinical validation of S100B in the management of a mild traumatic brain injury: issues from an interventional cohort of 1449 adult patients. Clin Chem Lab Med. 2018 Oct 25;56(11):1897-1904. doi: 10.1515/cclm-2018-0471. PMID 29924734
- [Background] Biberthaler P, Linsenmeier U, Pfeifer KJ, Kroetz M, Mussack T, Kanz KG, Hoecherl EF, Jonas F, Marzi I, Leucht P, Jochum M, Mutschler W. Serum S-100B concentration provides additional information fot the indication of computed tomography in patients after minor head injury: a prospective multicenter study. Shock. 2006 May;25(5):446-53. doi: 10.1097/01.shk.0000209534.61058.35. PMID 16680008
- [Background] Bouvier D, Oddoze C, Ben Haim D, Moustafa F, Legrand A, Alazia M, Jehle E, Schmidt J, Sapin V. [Interest of S100B protein blood level determination for the management of patients with minor head trauma]. Ann Biol Clin (Paris). 2009 Jul-Aug;67(4):425-31. doi: 10.1684/abc.2009.0347. French. PMID 19654082
- [Background] Calcagnile O, Unden L, Unden J. Clinical validation of S100B use in management of mild head injury. BMC Emerg Med. 2012 Oct 27;12:13. doi: 10.1186/1471-227X-12-13. PMID 23102492